CLINICAL TRIAL: NCT03900208
Title: The Arrhythmogenic Right Ventricular Cardiomyopathy/Dysplasia From Real World Autoptic Data: Diagnosis in the Absence of Clinical Criteria
Brief Title: The Arrhythmogenic Right Ventricular Cardiomyopathy/Dysplasia
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, clinical professor, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI 28.03.2019
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Right Ventricle Abnormality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hystological analysis of ventricular tissue — Sections (4μm thick) will be stained with hematoxylin and eosin stain (H&E) for diagnosis. After diagnosis, sections of the representative heart tissue will be stained with a PicroSirius Red/Fast Green for fibrosis evaluation. All stained samples will be examined under digital and light microscope. Beside the location of adipose/fibrous tissue in the right or left ventricles and in the septum, seven high magnification fields (40x) will be evaluated in five regions of the myocardium.

SUMMARY:
The arrhythmogenic right ventricular cardiomyopathy, also known as arrhythmogenic right ventricular dysplasia (ARVC/D) is a rare myocardial disease with a prevalence estimated to range from 1 case on 5000 persons in the general population. It have a dominant genetic transmission characterized by alterations of desmosomial proteins and predominantly affects the right ventricle. The morphological alteration of the myocardium characterized by fibro-fatty substitution predisposes to arrhythmic events that can be fatal and cause death especially in young people and athletes. International guidelines provide a classification that includes clinical and histological criteria for diagnosis based on fibrous tissue substitution, percentage and right ventricle localization. Indeed, it is mainly affected the right ventricle but in some cases also the left ventricle result involved and the fatty tissue or fibro-fatty tissue with particular arrangement may affect the full-thickness wall are pathognomonic. Authors identified 10 cases of arrhythmogenic cardiomyopathy in forensic autopsy collocated in the 2003 to 2017, included 8 males and 2 females. Their age ranged from 16 to 45 years with an average age of 28.8±8.1 years. However, authors would like to demonstrate that with ARVC/D cannot be include only cases with increased fibrosis and exclusive localization to the right ventricle nor even cases with electrocardiographic alterations and other evident clinical criteria. Indeed, in the analyzed cases authors observed an amount of fibrosis often less than the percentage reported in the literature and an involvement not only of the right ventricle but also of the septum and associated sinister ventricular modifications. To this must be added that the cases of death did not have a sudden death of relatives in family history as described in guidelines and therefore this criterion is not reliable for the purpose of a classification.

DETAILED DESCRIPTION:
The arrhythmogenic right ventricular cardiomyopathy/dysplasia (ARVC/D), have a prevalence estimated that range from 1 case on 5000 subjects in the general population to 1 in 2000 in some European countries such as Italy and Germany. It is a rare myocardial disease, with a dominant genetic transmission characterized by alterations of desmosomial proteins including desmoplakin (DSP), plakophilin 2 (PKP2), desmoglein 2 (DSG2), and desmocollin 2 (DSC2). ARVC/D mainly affects the right ventricle but in some cases also the left ventricle result involved and the fatty tissue or fibro-fatty tissue with particular arrangement may affect the full-thickness wall are pathognomonic. Progressive loss of right ventricular myocardium and its replacement by fibro-fatty tissue is the pathological hallmark of the disease and predisposes to the early onset of arrhythmias and sudden death especially in young people and athletes. The diagnosis is difficult and based on clinical major/minor criteria, including histological aspects based on fibrous tissue substitution (in percentage) and right ventricle localization. The introduction of the new term "borderline" ARVC allows to inform those individuals with undefined diseases for minor abnormalities that are at risk and require regular follow-up.

The histological criteria consist on microscopic observation of seven fields in five areas of the myocardium at a high magnification (40x) with the support of histochemical stains for the fibrous connective tissue and for the adipose tissue. Several studies have attempted to quantify the presence of adipose and fibrous tissue in the myocardial wall, and the value for histological diagnosis of ARVC provides a minimum 3% of adipose tissue and more than 40% of fibrous tissue. Conversely, other authors have suggested that a percentage of adipose tissue ranging from 5 to 20% is suspicious. This approach had limitations due to the lack of sensitivity of many of the criteria. Particularly, in ARVC families disease-causing mutation carriers often have very insidious results that do not usually lead to a diagnosis of ARVC in clinical practice. However, in te present research authors would demonstrated that with ARVC/D cannot be included only cases with increased fibrosis and exclusive localization to the right ventricle nor even cases with electrocardiographic alterations and other evident clinical criteria. The primary study goal of reviewing the guidelines will be reducing the dependence on subjective criteria to evaluate ventricular structure and function and to incorporating cardiac magnetic resonance and genetic analysis data. In the new system, patients should be diagnosed with "defined" ARVC if they have two major criteria, 1 major and 2 minor criteria, or 4 minor criteria of different categories and "borderline" ARVC with 1 major and 1 minor criteria, or 3 minors of different categories.

Materials and methods Patients and samples Authors will assay heart sections from 10 fatal cases of death, with an average age of 28.8±8.1 years (age ranged from 16 to 45 years), defined according to commonly accepted criteria and collected from January 2003 to December 2017 at the University of Naples Federico II. All the autopsies will be performed according to the Guidelines for autopsy investigation developed by the Association for European Cardiovascular Pathology, and in all cases they will be completely examined by macroscopic autopsy.

Histological evaluation In all cases, the sampling of ventricles, atria and septum including conduction system for the heart will be performed. The original tissues samples will be fixed in 10% neutral buffered formalin and embedded in paraffin blocks. Sections (4μm thick) will be stained with hematoxylin and eosin stain (H&E) for diagnosis. After diagnosis, sections of the representative heart tissue will be stained with a PicroSirius Red/Fast Green for fibrosis evaluation. All stained samples will be examined under digital and light microscope. Beside the location of adipose/fibrous tissue in the right or left ventricles and in the septum, seven high magnification fields (40x) will be evaluated in five regions of the myocardium.

ELIGIBILITY:
Inclusion Criteria:

* fatal cases of cardiac deaths
* both sexes
* aged more than 18 years and less than 75 years.

Exclusion Criteria:

* aged less than 18 years and more than 75 years
* patients without hystological diagnosis of right ventricle dysplasia.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population of bot sexes subjetcs aged more than 18 and less than 75 years, with diagnosis of right ventricle dysplasia (RVD), and linked worse prognosis with clinicla event of fatal death. All patients will receive an autopsy and an histopathological diagnosis of RVD as major study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
To measure the degree of fibrotic/fatty tissue alterations of right ventricle in patients with sudden unexplained death diagnosis. | 12 months
  Authors will measure the percentage of fibrotic/fatty tissue alterations of right ventricle from human samples .

IPD SHARING:
Plan to Share IPD: Undecided